CLINICAL TRIAL: NCT05686343
Title: Hemodynamically Important PDA in Newborns Under 32 Weeks: Clinical and Echocardiographic Findings and Outcomes
Brief Title: Hemodynamically Important Patent Ductus Arteriosus in Newborns Under 32 Weeks
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Özlem Bayram, Principal Investigator, Ankara University
Other Study IDs: Ankara University-001
Record Dates: First submitted 2022-12-26; First posted 2023-01-17 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2022-12

CONDITIONS: Patent Ductus Arteriosus After Premature Birth
Keywords: Cardiology; Newborn; Diseases; Congenital Heart Defects; Patent Ductus Arteriosus
MeSH Terms: conditions — Disease; Heart Defects, Congenital; Ductus Arteriosus, Patent | interventions — Echocardiography; Ultrasonography, Doppler; Spectroscopy, Near-Infrared

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Treated
  Interventions: Diagnostic Test: Echocardiography, Doppler ultrasonography, Near-infrared spectroscopy
- Untreated
  Interventions: Diagnostic Test: Echocardiography, Doppler ultrasonography, Near-infrared spectroscopy

INTERVENTIONS:
Diagnostic Test: Echocardiography, Doppler ultrasonography, Near-infrared spectroscopy — Ecocardiography at 1st, 3rd and 7th day of life Doppler US (cranial and renal) at 1st, 3rd and 7th day of life Near-infrared spectroscopy monitoring after birth during first 3-days of life

SUMMARY:
To define the characteristics of hemodynamically significant PDA by echocardiography, to investigate the systemic effects of the ductus with cerebral and renal Doppler flow studies, and to determine the oxygen consumption in the cerebral tissue with NIRS in newborns below 32 weeks of age with PDA.

ELIGIBILITY:
Inclusion Criteria:

* Born at less than 32 weeks newborns

Exclusion Criteria:

* Congenital heart disease
* Syndromic and/or major congenital anomaly

Ages: 1 Minute to 7 Days | Sex: All
Age Groups: Child
Study Population: Newborns < 32 weeks
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Diameter of PDA | 1 year
  Measurement the diameter of ductus in mm/weight using echocardiography
Velosity of PDA | 1 year
  Measurement the velosity of ductus using CW doppler on ecocardiyograpy
Left ventricule expansion | 1 year
  Measurement left ventricule end diastolic and end systolic diameter, left atrium/aort ratio on ecocardiography
Velocity of internal carotid arteries, middle carotid arteries, anterior cerebral arteries and renal arteries | 1 year
  Measurement velocity of internal carotid arteries, middle carotid arteries, anterior cerebral arteries and renal arteries using doppler ultrasonography

CONTACTS AND LOCATIONS:
Overall Officials: Özlem Bayram, Principal Investigator — Ankara University
Locations (1):
- Özlem Bayram, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No